CLINICAL TRIAL: NCT01159067
Title: Deferasirox Treatment and Labile Plasma Iron in Iron Overloaded Patients Who Have Undergone Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Deferasirox for Treating Patients Who Have Undergone Allogeneic Stem Cell Transplant and Have Iron Overload
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09187; NCI-2010-01428
Record Dates: First submitted 2010-07-06; First posted 2010-07-09 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2017-11

CONDITIONS: Iron Overload; Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Disseminated Neuroblastoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Poor Prognosis Metastatic Gestational Trophoblastic Tumor; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Neuroblastoma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage II Ovarian Epithelial Cancer; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Malignant Testicular Germ Cell Tumor; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Ovarian Epithelial Cancer; Stage III Small Lymphocytic Lymphoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Breast Cancer; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Ovarian Epithelial Cancer; Stage IV Small Lymphocytic Lymphoma
Keywords: HSCT, iron overload, deferasirox, labile plasma iron
MeSH Terms: conditions — Iron Overload; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Testicular Neoplasms; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral deferasirox once daily for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox — Given orally
  Other Names: Exjade; ICL670

SUMMARY:
RATIONALE: Low dose deferasirox may be safe and effective in treating patients who have undergone hematopoietic stem cell transplant and have iron overload.

PURPOSE: This pilot clinical trial studies safety and tolerability of deferasirox in hematopoietic stem cell transplant recipients who have iron overload. Effect of low dose deferasirox on labile plasma iron is also examined.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine labile plasma iron (LPI) levels in iron overloaded patients after allogeneic Hematopoietic Stem Cell Transplantation (HSCT).

II. To determine safety and tolerability of low dose deferasirox in the post allogeneic HSCT setting.

SECONDARY OBJECTIVES:

I. To determine ability of deferasirox to suppress LPI in allogeneic HSCT patients with serum ferritin over 1500 ng/ml.

II. To determine prevalence of elevated LPI in allogeneic HSCT recipients with serum ferritin over 1500 ng/ml.

III. To determine ability of low dose deferasirox to lower serum ferritin during the treatment period.

IV. To correlate LPI with serum ferritin in allogeneic HSCT recipients with serum ferritin over 1500 ng/ml.

OUTLINE: Patients receive deferasirox at 10 mg/kg once daily for 6 months in the absence of unacceptable toxicity. Labile plasma iron will be measured at baseline and at weeks 4, 12, and 24. Side effects of deferasirox will be recorded.

ELIGIBILITY:
Inclusion

* Patients must have undergone a matched related donor, matched unrelated donor or cord blood Hematopoietic Stem Cell Transplant (HSCT) over 6 months ago
* Patients currently on Desferal (desferrioxamine) therapy will require a one day wash out prior to the first dose of study drug
* Serum ferritin >= 1500 ng/mL on two occasions two weeks apart at screening; samples must be obtained in the absence of concomitant infection
* Normal C-reactive protein level at screening
* Patients must be red cell transfusion independent for 2 months prior to enrollment
* Sexually active women must use an effective method of contraception, or must have undergone clinical documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal (defined as amenorrhea for at least 12 months)
* Written informed consent by the patient

Exclusion

* Chronic hepatic GVHD with serum total bilirubin over 2 mg/dL
* Known hypersensitivity to deferasirox
* Serum creatinine above the upper limit of normal
* AST or ALT > 200 U/L during screening
* Clinical or laboratory evidence of active Hepatitis B or Hepatitis C (HBsAg in the absence of HBsAb OR HCV Ab positive with HCV RNA positive and ALT above the normal range)
* History of HIV positive test result (ELISA or Western blot)
* History of drug or alcohol abuse within the 12 months prior to enrollment
* ECOG Performance Status > 2
* Patients with a diagnosis of or history of clinically relevant ocular toxicity related to iron chelation
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent study treatment
* Pregnancy (as documented in required screening laboratory test) or breast feeding
* Patients who received treatment with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days or are planning to receive other investigational drugs while participating in the study
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug
* History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08-09 (Actual); Study Completion 2011-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Pullarkat, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Elevated Labile Plasma Iron (LPI) Above Threshold (0.5 Umol/L)
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Number of Patients With LPI Below 0.5 Umol/L After Treatment
Description: In patients with LPI values above threshold 0.5umol/L at baseline, number of patients had LPI suppressed below this value after treatment. Measurement of LPI is done on plasma specimens.
Time Frame: Assessed through 6 months from the start of treatment
Population: No patient had elevated LPI level above 0.5umol/L at baseline.
Arm/Group | Arm I
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With Serum Ferritin Level Lower Than 1500 ng/mL After Treatment
Description: Number of patients, whose Serum Ferritin levels are lower than 1500 ng/mL at two consecutive study visits. Serum Ferritin levels are measured at screening (baseline), week 4, 8, 12, 16, 20, 24 and end of study.
Time Frame: Assessed through 6 months from the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Correlation of LPI With Serum Ferritin
Description: Both LPI and Serum Ferritin levels are measured at screening (baseline), week 4, 12, 24 and end of study. The correlation between the levels of LPI and Serum Ferritin at screening, week 4, 12, 24 and end of study will be examined and plotted.
Time Frame: Assessed through 6 months from the start of treatment
Population: The enrolled patient's LPI level at baseline is below 0.5 umol/L and she had both LPI and Serum Ferritin levels measured at baseline only. Therefore, no sufficient data to estimate the correlation of LPI with Serum Ferritin.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Cycle 1 to Cycle 6
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=1)
Iron overload (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (2)
Platelets (Blood and lymphatic system disorders) | 1 (10)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Fever (General disorders) | 1 (1) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Rigors/chills (General disorders) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (6)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (6)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU (Gastrointestinal disorders) | 1 (5)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 1 (2) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (6)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (6)
Creatinine (Metabolism and nutrition disorders) | 1 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (3)
Proteinuria (Metabolism and nutrition disorders) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes